CLINICAL TRIAL: NCT07083752
Title: Investigation of the Effects of Upper Extremity Botulinum Toxin Application on Forearm Muscle Thickness and Motor Recovery in Patients With Hemiplegia
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, assistant professor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-SK-10
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hemiplegia; Spasticity, Muscle
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Botulinum toxin application — Hemiplegic stroke patients who received upper extremity botulinum toxin will be evaluated retrospectively. Information regarding upper extremity motor recovery, spasticity levels, and muscle thickness measured by ultrasound before and one month after botulinum toxin administration will be obtained from file records.

SUMMARY:
In this study, we aimed to examine the effects of the botulinum toxin (BoNT) application on muscle thickness and motor recovery in stroke patients.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death worldwide. It poses a major risk for disability. Its prevalence is high in developing countries. Spasticity is among the complications of stroke. Excessive spasticity can cause impairments and limitations in patients' motor activity and participation in daily life. Botulinum toxin (BoNT) injection is one of the preferred treatment options. Studies on botulinum toxin administration in stroke patients generally focus on treatment efficacy and motor recovery. Studies examining the effects of botulinum toxin administration on both muscle thickness and motor recovery are few in number. In this study, we aimed to examine the effects of the botulinum toxin (BoNT) application on upper extremity muscle thickness and motor recovery in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between the ages of 30-75.
* Patients who received botulinum toxin injection to their upper extremities at least 3 months after a cerebrovascular accident.
* Patients must have had cerebrovascular disease for the first time.

Exclusion Criteria:

* Presence of a preexisting musculoskeletal deformity in the upper extremity where botulinum toxin was administered
* Patients with spinal cord injury, multiple sclerosis, and cerebral palsy
* Presence of malignancy.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was designed as a retrospective cross-sectional study. The study included patients who had been hospitalized at İzzet Baysal Physical Therapy and Rehabilitation Education and Research Hospital with a diagnosis of hemiplegia due to stroke, had participated in a rehabilitation program, had given informed consent previously, and had received botulinum toxin injections to their upper extremities.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-07-13 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Muscle Thickness | Before treatment
  Muscle thickness measurements were performed using a Falcon 2101 EXL 2003 ultrasound device equipped with an 8 MHz linear probe, both before and one month after botulinum toxin application.
  In patients who received botulinum toxin injections into the m. brachialis, m. pronator teres, m. flexor carpi radialis, m. flexor carpi ulnaris, m. flexor digitorum profundus, and m. flexor digitorum superficialis, muscle thickness was measured using ultrasound from the proximal one-third of the volar side of the forearm. Measurements were taken before and one month after the application. Muscle thickness was recorded by measuring the vertical distance between the subcutaneous tissue and the radius and ulna bone borders on the ultrasound image.
Muscle Thickness | 4 week after treatment
  Muscle thickness measurements were performed using a Falcon 2101 EXL 2003 ultrasound device equipped with an 8 MHz linear probe, both before and one month after botulinum toxin application.
  In patients who received botulinum toxin injections into the m. brachialis, m. pronator teres, m. flexor carpi radialis, m. flexor carpi ulnaris, m. flexor digitorum profundus, and m. flexor digitorum superficialis, muscle thickness was measured using ultrasound from the proximal one-third of the volar side of the forearm. Measurements were taken before and one month after the application. Muscle thickness was recorded by measuring the vertical distance between the subcutaneous tissue and the radius and ulna bone borders on the ultrasound image.
Brunnstrom Motor Recovery Stages | Before treatment
  Brunnstrom stages is a scale used to assess motor recovery after a stroke, which is expressed using values between 1 and 6. The higher the value on this scale, the higher would be the recovery.
Brunnstrom Motor Recovery Stages | 4 week after treatment
  Brunnstrom stages is a scale used to assess motor recovery after a stroke, which is expressed using values between 1 and 6. The higher the value on this scale, the higher would be the recovery.

SECONDARY OUTCOMES:
Modified Ashworth Scale | Before treatment
  Spasticity in the shoulder will be evaluated according to the Modified Ashworth Scale (MAS). The Modified Ashworth Scale is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent increased degree of spasticity.
Modified Ashworth Scale | 4 week after treatment
  Spasticity in the shoulder will be evaluated according to the Modified Ashworth Scale (MAS). The Modified Ashworth Scale is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent increased degree of spasticity.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No